CLINICAL TRIAL: NCT06129214
Title: Partial Synovectomy in Articular Side of Quadriceps Tendon Reduces Crepitus After Posterior Stabilized Total Knee Arthroplasty : a Randomized, Controlled Trial
Brief Title: Partial Synovectomy in Articular Side of Quadriceps Tendon Verified to Reduce Crepitus in Retrospective Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Woo Suk Lee, professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2023-0282
Record Dates: First submitted 2023-10-18; First posted 2023-11-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis, Knee; Spontaneous Osteonecrosis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synovium removal group (Experimental)
  Interventions: Procedure: Prepectoral; Procedure: Subpectoral
- Synovium sustain group (No Intervention)

INTERVENTIONS:
Procedure: Prepectoral — Remove all visible synovium in suprapatellar area under distal quadriceps tendon. All other procedures (Total Knee arthroplasty) are same with no intervention arm.
  Arms: Synovium removal group
Procedure: Subpectoral — No remove any synovium in suparapatellar area under distal quadriceps tendon. All other preocedures are same with experimental arm.
  Arms: Synovium removal group

SUMMARY:
Crepitus causing unsatisfied result to patients after posterior stabilized total knee arthroplasty. Recent retrospective study demonstrated removal of hyperplastic synovium in distal quadriceps caused reduce of crepitus. However, this study has limitation of time gap exist between arms, different in observation time and bias caused by retrospective review. Thus aim of this study is that by randomized trial, verified hyperplastic synovium in distal quadriceps causing crepitus.

Target enrolled patients in this study are scheduled to perform both total knee arthroplasty. Experimental group is randomized side (right or left) of knee, and control group is other side of knee. Both arms decided by randomized number table. Crepitus measured after 3mo, 6mo, 1year after surgical treatment

DETAILED DESCRIPTION:
Surgical treatment of TKA with synovium removal in distal quadriceps tendon performed classifed as experimental arm and TKA wiout synovium removal classified as control arm. Before surgical treatment, radiologic and physiological evaluation performed to check too much variance shown in either arm. Radiologic parameter include Hip knee ankle angle, Femoral tibial angle, Level of joint line, Insall-Salvati ratio, Posterior tibial slope, Posterior femoral condylar offset, Patellar thickness, Patellar tilt, Patellar displacement. During surgical treatment patella resurfacing in either group excluded this study. Indication of patella resufacing is ICRS grade IV in lateral surface of patella. After surgical procedure done check grade of crepitus (0-no crepitation, 1-fine crepitation, 2-coarse crepitation) with WOMAC, Knee Society Score, Eq-5D (European quality of life -5 Dimensions), Forgotten joint score after 3month, 6month and 1year after surgical procedure.

Other collecting variance Age, Gender, BMI, Range of motion of knee, Fmoeral/Tibial component size, PE thickness

ELIGIBILITY:
Inclusion Criteria:

1.Patients who scheduled to perform both total knee arthroplasty(TKA) using posteiror crucitate sustain type (PS)

Exclusion Criteria:

1. Lost follow up (Including death of patient)
2. Unexpected complication (e.g) Infection, periprosthetic fracture)
3. Patella resurfacing
4. Canceled surgical treatment
5. Refused to enrolled study
6. Too much radiological or physicological variance shown between either knee

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Crepitus grade | 3month, 6month, 1year after surgical treatment
  Crepitus grade divided 3 categories ; 0-no crepitus, 1-asymptomatic crepitus, 2-Painful crepitus

SECONDARY OUTCOMES:
Hip knee ankle angle | 3month, 6month, 1year after surgical treatment
  Identify postop alignment of lower extrimities, which is mechanical axis between femur and tibia in scanogram of low extremity.
Insall-Salvati ratio | 3month, 6month, 1year after surgical treatment
  Measured in true lateral position in 30' knee flextion, measureing patellar position in lateral plain radiograph of knee.
Patellar displacement | 3month, 6month, 1year after surgical treatment
  Measuring patellar position in merchant view of plain radiograph.
Patellar tilt angle | 3month, 6month, 1year after surgical treatment
  Measuring patellar position in merchant view of plain radiograph.
Tibia offset | 3month, 6month, 1year after surgical treatment
  Estimate tibial component position in lateral plain radiograph.
Knee society score | 3month, 6month, 1year after surgical treatment
  Clinical score evaluate functional ability of patients after surgery (0-100; high value represent better outcome)
WOMAC score | 3month, 6month, 1year after surgical treatment
  Clinical score evaluate pain, stiffness, function of knee after surgery (0-96; low value represent better outcome)
Forgotten joint score | 3month, 6month, 1year after surgical treatment
  Clinical score evaluate functional outcome after surgery (0-100; low value represent better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, GangnamGu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chumchuen S, Kanitnate S, Wattanasirisombat K, Tammachote N. Synovium removal from the articular side of the quadriceps tendon around the superior pole of patella reduces the crepitus after total knee arthroplasty. Int Orthop. 2022 Nov;46(11):2561-2567. doi: 10.1007/s00264-022-05539-2. Epub 2022 Aug 13. PMID 35962233